CLINICAL TRIAL: NCT05212727
Title: Development and Validation of a Novel Functional Eye-Tracking Software Application for Neurological Disorders
Status: Suspended | Type: Observational
Why Stopped: Insufficient personnel
Sponsor: Innodem Neurosciences (Industry)
Responsible Party: Sponsor
Other Study IDs: ETNA-NDHC
Record Dates: First submitted 2022-01-18; First posted 2022-01-28 (Actual); Last update posted 2024-03-05 (Actual); Status verified 2024-03

CONDITIONS: Neurological Disorders
Keywords: Neurological disorders; Eye-tracking; Eye Movement Biomarkers
MeSH Terms: conditions — Nervous System Diseases | interventions — Eye-Tracking Technology

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Healthy Control: Participant with no evidence or history of significant neurodegenerative disorder affecting brain function.
  Interventions: Device: Eye-tracking

INTERVENTIONS:
Device: Eye-tracking — Eye-tracking technology and algorithms used to successfully capture and track eye movements using an electronic tablet and the embedded camera of the device.

SUMMARY:
This study aims to develop and validate a sensitive and non-invasive eye-tracking software application.

This study will obtain participant responses to brief cognitive tests designed to evaluate several key functions known to be affected by neurological disorders and non-invasive eye movement measurements in response to visually presented stimuli during specifically designed eye-tracking tests. The study data will be used to develop machine learning algorithms and validate a software application intended to track the progressive component of neurological disorders and associated cognitive changes.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years old and above
* A score of ≥ 26 on the Montreal Cognitive Assessment (MoCA)
* Able to provide informed consent
* Visual acuity of 20/100 in at least one eye (corrective glasses, contact lenses, surgery etc are permitted).

Exclusion Criteria:

* Evidence or medical history of psychiatric issues, which are known to also affect movements and oculomotor control.
* Evidence or history of significant neurological disorder (e.g. MS, PD, ALS, Dementia)
* Use of prescription drugs known to influence ocular motor visual function, such as benzodiazepines, antipsychotics, and anticonvulsants.
* Diagnosed with an active substance use disorder.
* History of stroke.
* Recent traumatic brain injury (within the last 6 months).

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Data will be obtained from 300 healthy adult individuals across the age spectrum. We will stop recruiting participants of a certain age once one of the following age groups has reached 100 participants:
  18-40 40-60 60 and over
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2022-04-15 (Actual); Primary Completion 2024-05-03 (Estimated); Study Completion 2024-05-03 (Estimated)

PRIMARY OUTCOMES:
Symbol Digit Modalities Test (SDMT) score, one time, at the day of enrolment. | Baseline
  The SDMT is used to assess divided attention, visual scanning, tracking and motor speed. Using a reference key, the examinee has 90 seconds to pair specific numbers with given geometric figures. Scoring involves summing the number of correct substitutions within the 90 second interval.

SECONDARY OUTCOMES:
Brief International Cognitive Assessment for MS (BICAMS) score, one time, at the day of enrolment. | Baseline
  The BICAMS is a battery of tests recommended by multiple sclerosis (MS) experts to monitor MS-related cognitive impairment. It includes the Symbol Digit Modalities Test (SDMT), the California Verbal Learning Test-2 (CVLT2) and the Brief Visuospatial Memory Test-Revised (BVMT-R)
Multiple sclerosis functional composite (MSFC) score, one time, at the day of enrolment. | Baseline
  A clinical trial outcome measure of assessing the severity of multiple sclerosis (MS) primarily. used in research. The score is based on a combination of timed tests of walking, arm function, and cognitive ability. It is a three-part, standardized, quantitative, assessment instrument for use in clinical studies, particularly clinical trials, of MS. The MSFC can produce scores for each of the three individual measures as well as a composite score.
The Montreal Cognitive Assessment (MoCA) score, one time, at the day of enrolment. | Baseline
  The Montreal Cognitive Assessment (MoCA) is a brief 30-question cognitive screening test designed to assist Health Professionals in the detection of mild cognitive impairment and Alzheimer's disease. It assesses different cognitive domains: attention and concentration, executive functions, memory, language, visuoconstructional skills, conceptual thinking, calculations, and orientation.
  Scores on the MoCA range from zero to 30, with a score of 26 and higher generally considered normal.
The Mini-Mental State Exam (MMSE) score, one time, at the day of enrolment. | Baseline
  The Mini-Mental State Exam (MMSE) is a widely used test of cognitive function among the elderly, it includes tests of orientation, attention, memory, language and visual-spatial skills. It consists of a series of questions and tests that can be used by clinicians to help diagnose dementia and to help assess its progression and severity.
The Controlled Oral Word Association Test (COWAT) score, one time, at the day of enrolment. | Baseline
  The Controlled Oral Word Association Test from the Halstead-Reitan Neuropsychological Battery is a verbal fluency test in which participants are asked to say as many words as possible from a given category and in a specified timeframe (typically 60 seconds).
The Trail Making Test (TMT) Parts A & B score, one time, at the day of enrolment. | Baserline
  The Trail Making Test (TMT) is a neuropsychological test that provides information on visual search, scanning, speed of processing, mental flexibility and executive functions. The TMT consists of two parts. TMT-A requires an individual to draw lines sequentially connecting 25 encircled numbers distributed on a sheet of paper. Task requirements are similar for TMT-B except the person must alternate between numbers and letters (e.g., 1, A, 2, B, 3, C, etc.). The score on each part represents the amount of time required to complete the task.
The Hopkins Verbal Learning Test-Revised (HVLT-R) score, one time, at the day of enrolment. | Baseline
  The Hopkins Verbal Learning Test (HVLT-R) is a neuropsychological test that provides information on verbal learning and memory. The assessment consists of memorization of a list of words to test the ability to recall immediately after memorization (immediate recall) and after a 20-minute delay (delayed recall).
The Functional Assessment of Cancer Therapy - Cognitive Function (FACT-Cog), one time, at the day of enrolment. | Baseline
  The Functional Assessment of Cancer Therapy-Cognitive Function (FACT-Cog), currently in its third version, is a questionnaire that evaluates patients' self-reported perceptions of their cognitive abilities and the effects of these cognitive changes on their Health-related quality of life (HRQOL).
The Beck Anxiety Inventory (BAI), one time at the day of enrolment. | Baseline
  The Beck Anxiety Inventory (BAI) consists of 21 self-reported items (four-point scale) used to assess the intensity of physical and cognitive anxiety symptoms during the past week. Scores may range from 0 to 63: minimal anxiety levels (0-7), mild anxiety (8-15), moderate anxiety (16-25), and severe anxiety (26-63).

CONTACTS AND LOCATIONS:
Locations (1):
- Innodem Neurosciences, Montreal, Quebec, Canada